CLINICAL TRIAL: NCT02161718
Title: A Phase 2, Efficacy, Safety and Tolerability Study of ALKS 3831 in Schizophrenia With Alcohol Use Disorder
Brief Title: A Study of ALKS 3831 in Subjects With Schizophrenia and Alcohol Use Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alkermes, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALK3831-401
Record Dates: First submitted 2014-05-28; First posted 2014-06-12 (Estimated); Results first posted 2021-10-08 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2021-09

CONDITIONS: Schizophrenia; Alcohol Use Disorder
Keywords: Alkermes; Schizophrenia; Alcohol Use Disorder; ALKS 3831
MeSH Terms: conditions — Schizophrenia; Alcoholism | interventions — 3-carboxamido-4-hydroxynaltrexone; Olanzapine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Samidorphan + olanzapine (ALKS 3831) (Experimental): Active study drug
  Interventions: Drug: Samidorphan + olanzapine (ALKS 3831)
- Placebo + olanzapine (Placebo Comparator)
  Interventions: Drug: Placebo + olanzapine

INTERVENTIONS:
Drug: Samidorphan + olanzapine (ALKS 3831) — Oral tablet, taken once daily
  Arms: Samidorphan + olanzapine (ALKS 3831)
Drug: Placebo + olanzapine — Oral tablet, taken once daily
  Arms: Placebo + olanzapine

SUMMARY:
This double-blind, randomized study will evaluate the efficacy, safety and tolerability of ALKS 3831 in subjects with schizophrenia and alcohol use disorder (AUD).

ELIGIBILITY:
Inclusion Criteria:

* Has a BMI between 18.0 and 40.0 kg/m2, inclusive
* Has a diagnosis of schizophrenia
* Has a diagnosis of alcohol use disorder (AUD)
* Has experienced an acute exacerbation of schizophrenia within the past 6 months
* Additional criteria may apply

Exclusion Criteria:

* Is pregnant or breastfeeding
* Had first lifetime psychotic episode less than 1 year before screening or has experienced only a single lifetime psychotic episode
* Has a known or suspected intolerance, allergy, or hypersensitivity to olanzapine
* Has current or pending legal charges with the potential for incarceration
* Has a positive drug screen for opiates
* Additional criteria may apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2017-01-11 (Actual); Study Completion 2017-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David McDonnell, MD, Study Director — Alkermes, Inc.
Locations (65):
- United States (53):
  - Alkermes Investigational Site, Little Rock, Arkansas
  - Alkermes Investigational Site, Springdale, Arkansas
  - Alkermes Investigational Site, Anaheim, California
  - Alkermes Investigational Site, Culver City, California
  - Alkermes Investigational Site, Garden Grove, California
  - Alkermes Investigational Site, Irvine, California
  - Alkermes Investigational Site, La Jolla, California
  - Alkermes Investigational Site, Long Beach, California
  - Alkermes Investigational Site, National City, California
  - Alkermes Investigational Site, Oakland, California
  - Alkermes Investigational Site, Oceanside, California
  - Alkermes Investigational Site, Orange, California
  - Alkermes Investigational Site, San Diego, California
  - Alkermes Investigational Site, San Francisco, California
  - Alkermes Investigational Site, Torrance, California
  - Alkermes Investigational Site, Washington D.C., District of Columbia
  - Alkermes Investigational Site, Fort Lauderdale, Florida
  - Alkermes Investigational Site, Leesburg, Florida
  - Alkermes Investigational Site, Maitland, Florida
  - Alkermes Investigational Site, Miami, Florida
  - Alkermes Investigational Site, North Miami, Florida
  - Alkermes Investigational Site, Oakland Park, Florida
  - Alkermes Investigational Site, Orlando, Florida
  - Alkermes Investigational Site, Tampa, Florida
  - Alkermes Investigational Site, Atlanta, Georgia
  - Alkermes Investigational Site, Augusta, Georgia
  - Alkermes Investigational Site, Decatur, Georgia
  - Alkermes Investigational Site, Chicago, Illinois
  - Alkermes Investigational Site, Hoffman Estates, Illinois
  - Alkermes Investigational Site, Oak Brook, Illinois
  - Alkermes Investigational Site, Shreveport, Louisiana
  - Alkermes Investigational Site, Worcester, Massachusetts
  - Alkermes Investigational Site, Flowood, Mississippi
  - Alkermes Investigational Site, Creve Coeur, Missouri
  - Alkermes Investigational Site, Kansas City, Missouri
  - Alkermes Investigational Site, St Louis, Missouri
  - Alkermes Investigational Site, Las Vegas, Nevada
  - Alkermes Investigational Site, Claremont, New Hampshire
  - Alkermes Investigational Site, Nashua, New Hampshire
  - Alkermes Investigational Site, Neptune City, New Jersey
  - Alkermes Investigational Site, Cedarhurst, New York
  - Alkermes Investigational Site, Jamaica, New York
  - Alkermes Investigational Site, New York, New York
  - Alkermes Investigational Site, Rochester, New York
  - Alkermes Investigational Site, Staten Island, New York
  - Alkermes Investigational Site, Dayton, Ohio
  - Alkermes Investigational Site, Oklahoma City, Oklahoma
  - Alkermes Investigational Site, Scranton, Pennsylvania
  - Alkermes Investigational Site, Charleston, South Carolina
  - Alkermes Investigational Site, Austin, Texas
  - Alkermes Investigational Site, Dallas, Texas
  - Alkermes Investigational Site, DeSoto, Texas
  - Alkermes Investigational Site, Bellevue, Washington
- Bulgaria (8):
  - Alkermes Investigational Site, Burgas
  - Alkermes Investigational Site, Kazanlak
  - Alkermes Investigational Site, Lovech
  - Alkermes Investigational Site, Novi Iskar
  - Alkermes Investigational Site, Sofia
  - Alkermes Investigational Site, Tserova Koria
  - Alkermes Investigational Site, Varna
  - Alkermes Investigational Site, Vratsa
- Poland (4):
  - Alkermes Investigational Site, Bełchatów
  - Alkermes Investigational Site, Bialystok
  - Alkermes Investigational Site, Gdansk
  - Alkermes Investigational Site, Lublin

REFERENCES:
- [Result] Brunette MF, Correll CU, O'Malley SS, McDonnell D, DiPetrillo L, Jiang Y, Simmons A, Silverman BL, Citrome L, Green AI. Olanzapine Plus Samidorphan (ALKS 3831) in Schizophrenia and Comorbid Alcohol Use Disorder: A Phase 2, Randomized Clinical Trial. J Clin Psychiatry. 2020 Mar 10;81(2):19m12786. doi: 10.4088/JCP.19m12786. PMID 32160422

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were adults with a diagnosis of schizophrenia and Alcohol Use Disorder (AUD). Subjects must also have recently experienced an exacerbation of disease symptoms (eg, hospitalization), but could not exceed a pre-defined level of symptom severity at the time of screening (as measured by assessments like the Positive and Negative Symptom Scale [PANSS] and Clinical Global Impression- Severity [CGI-S]).
Pre-assignment Details: After screening, subjects began a 4-week open-label olanzapine dosing period followed by a 2- week open-label ALKS 3831 period. Subjects who did not tolerate ALKS 3831 during the second open-label period were discontinued from the study prior to randomization. A total of 300 subjects were enrolled in the study, and 255 completed the open-label olanzapine period. 234 subjects were randomized following the open-label ALKS 3831 period, however, 5 subjects discontinued prior to receiving treatment.
Groups:
- Open-label ALKS 3831; ALKS 3831: Oral tablet, taken once daily ALKS 3831: Olanzapine (dose level determined by investigator) + Samidorphan (10mg)
- Olanzapine + Placebo: Oral tablet, taken once daily
  Olanzapine dose level determined by investigator
Period: Open-Label ALKS 3831 Period
Arm/Group | Open-label ALKS 3831 | ALKS 3831 | Olanzapine + Placebo
Started | 255 | 0 | 0
Completed | 234 | 0 | 0
Not Completed | 21 | 0 | 0
Not completed — Protocol Violation | 2 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0
Not completed — Non-compliance with study drug | 1 | 0 | 0
Not completed — Lack of Efficacy | 1 | 0 | 0
Not completed — Adverse Event | 3 | 0 | 0
Not completed — Withdrawal by Subject | 4 | 0 | 0
Not completed — Lost to Follow-up | 3 | 0 | 0
Not completed — Failure to meet randomization criteria | 6 | 0 | 0
Period: Post- Randomization Period
Arm/Group | Open-label ALKS 3831 | ALKS 3831 | Olanzapine + Placebo
Started | 0 | 112 | 117
Completed | 0 | 53 | 58
Not Completed | 0 | 59 | 59
Not completed — Withdrawal by Subject | 0 | 23 | 18
Not completed — Lost to Follow-up | 0 | 9 | 15
Not completed — Adverse Event | 0 | 9 | 10
Not completed — Non- compliance with study drug | 0 | 8 | 2
Not completed — Physician Decision | 0 | 2 | 4
Not completed — Protocol Violation | 0 | 2 | 3
Not completed — Lack of Efficacy | 0 | 0 | 1
Not completed — Non-compliance with study procedures | 0 | 2 | 4
Not completed — Received prohibitive treatment | 0 | 1 | 2
Not completed — Relocation | 0 | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ALKS 3831 | Olanzapine + Placebo | Total
Number analyzed (Participants) | 112 | 117 | 229
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.4 (10.60) | 45.1 (10.22) | 45.7 (10.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 26 | 49
  Male | 89 | 91 | 180
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 7 | 11
  Not Hispanic or Latino | 108 | 109 | 217
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 2
  Black or African American | 65 | 57 | 122
  White | 43 | 58 | 101
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 85 | 76 | 161
  Bulgaria | 24 | 36 | 60
  Poland | 3 | 5 | 8
Height [Mean (Standard Deviation); unit: centimeters] | 173.4 (9.6) | 174.4 (8.4) | 173.9 (9.0)
Weight [Mean (Standard Deviation); unit: kilograms] | 86.2 (19.7) | 86.8 (18.1) | 86.5 (18.9)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 28.6 (5.7) | 28.5 (5.4) | 28.6 (5.6)
Body Mass Index (BMI) Group [Count of Participants; unit: Participants]
  Underweight (<18.5) | 3 | 0 | 3
  Normal (18.5 to <25) | 34 | 29 | 63
  Overweight (25 to <30) | 33 | 49 | 82
  Obese (>= 30) | 42 | 39 | 81

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Independent Adjudication Committee (IAC) Adjudicated Event of Exacerbation of Disease (EEDS)
Description: EEDS was defined as any of the following occurring during the double-blind period & was related to worsening of disease symptoms, as confirmed by the Independent Adjudication Committee (IAC):
  1. Hospitalization (includes psychiatric& treatment of alcohol intoxication/withdrawal)
  2. >= 25% or >= 15 point increase from randomization in PANSS total score
  3. PANSS items score of P1, P2, P3, P6, P7 or G8 that meets 1 of the following:
  3a. Score >= 5 for subjects at a 2nd ad hoc visit with a score <=3 at randomization 3b. Score >= 6 for subjects at a 2nd ad hoc visit with a score =4 at randomization 4. Engagement in self injury, aggressive behavior, or suicidal/homicidal ideation 5. Initiation of rescue medication, including increase in olanzapine dosage initially prescribed at randomization 6. ER visit 7. Subject withdraws or PI discontinues subject for lack of efficacy, lost to follow-up, or withdrawal by subject 8. Arrest or incarceration related to subject's underlying disease
Time Frame: Up to 15 months
Population: Efficacy analyses were carried out using the intent to treat (ITT) population, i.e. all randomized subjects who received at least one dose of study drug post-randomization
Measure: Count of Participants; unit: Participants
Arm/Group | ALKS 3831 | Olanzapine + Placebo
Number analyzed (Participants) | 112 | 117
Participants
  Number of Subjects with IAC Adjudicated EEDS | 25 | 29
  Number of Subjects Censored | 87 | 88
Statistical Analysis 1: Comparison: ALKS 3831 vs Olanzapine + Placebo; Test type: Superiority; p = 0.746, Log Rank; Hazard Ratio (HR) = 0.91, 95% CI 2-sided [0.53 to 1.56], Standard Error of Mean 0.251

2. Secondary Outcome: Number of Events of Exacerbation of Disease (EEDS)
Description: EEDS was defined as any of the following occurring during the double-blind period & was related to worsening of disease symptoms, as confirmed by the Independent Adjudication Committee (IAC):
  1. Hospitalization(includes psychiatric & treatment of alcohol intoxication/withdrawal)
  2. >= 25% or >= 15 point increase from randomization in PANSS total score
  3. PANSS items score of P1, P2, P3, P6, P7 or G8 that meets 1 of the following:
  3a. Score >= 5 for subjects at a 2nd ad hoc visit with a score <=3 at randomization 3b. Score >= 6 for subjects at a 2nd ad hoc visit with a score =4 at randomization 4. Engagement in self injury, aggressive behavior, or suicidal/homicidal ideation 5. Initiation of rescue medication, including increase in olanzapine dosage initially prescribed at randomization 6. ER visit 7. Subject withdraws or PI discontinues subject for lack of efficacy, lost to follow-up, or withdrawal by subject 8. Arrest or incarceration related to subject's underlying disease
Time Frame: Up to 15 months
Population: as for outcome 1
Measure: Number; unit: Events
Arm/Group | ALKS 3831 | Olanzapine + Placebo
Number analyzed (Participants) | 112 | 117
Events | 35 | 49
Statistical Analysis 1: Comparison: ALKS 3831 vs Olanzapine + Placebo; Test type: Superiority; p = 0.372, Andersen-Gill Recurrent-Event Cox Model; Hazard Ratio (HR) = 0.77, 95% CI 2-sided [0.43 to 1.37]

3. Secondary Outcome: Number and Percentage of Subjects With at Least 1 Level Decrease in World Health Organization (WHO) Drinking Risk Level From Baseline to Week 24 of the Double-blind Treatment (Study Week 27)
Description: Alcohol consumption per day = (total number of drinks x 14 gram) / (total number of days)
  WHO criteria for risk of alcohol consumption on a single drinking day:
  Abstinence- Males: 0 g; Females- 0 g Low Risk- Males: 1-40 g; Females: 1-20 g Medium Risk- Males: 41- 60 g; Females: 21- 40 g High Risk- Males: 61-100 g; Females: 41-60 g Very High Risk- Males: >= 101 g; Females: >= 61 g
Time Frame: 24 weeks
Population: Efficacy analyses were carried out using subjects from the intent to treat (ITT) population with postbaseline data on drinking habits.
Measure: Count of Participants; unit: Participants
Arm/Group | ALKS 3831 | Olanzapine + Placebo
Number analyzed (Participants) | 111 | 116
Participants
  >= 1 Level Decrease from Baseline | 45 | 44
  < 1 Level Decrease from Baseline | 66 | 72
Statistical Analysis 1: Comparison: ALKS 3831 vs Olanzapine + Placebo; Test type: Superiority; p = 0.963, Regression, Logistic; Odds Ratio (OR) = 0.99, 95% CI 2-sided [0.56 to 1.73]

ADVERSE EVENTS:
Time Frame: Adverse events are presented for the randomized, double-blind period (9-15 months) as well as the 2 week open-label ALKS 3831 (olanzapine + samidorphan) period for a total timeframe of up to 62 weeks.
Groups:
- Open- Label ALKS 3831: A 2-week open-label period; all subjects received olanzapine (dose determined by investigator) + 10 mg samidorphan
- Olanzapine + Placebo: All randomized subjects who received at least 1 dose of study drug (olanzapine + placebo) during the double-blind treatment period
- ALKS 3831: All randomized subjects who received at least 1 dose of ALKS 3831 (olanzapine + samidorphan) during the double-blind treatment period.
Arm/Group | Open- Label ALKS 3831 | Olanzapine + Placebo | ALKS 3831
All-Cause Mortality (participants affected / at risk) | 0/255 | 1/117 | 1/112
Serious Adverse Events (participants affected / at risk) | 4/255 | 12/117 | 7/112
Other Adverse Events (participants affected / at risk) | 0/255 | 19/117 | 26/112
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Open- Label ALKS 3831 (N=255) | Olanzapine + Placebo (N=117) | ALKS 3831 (N=112)
Parotitis (Infections and infestations) | 0 | 1 | 0
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0
Electrocardiogram abnormal (Investigations) | 0 | 0 | 1
Chronic obstructive pulmonary disease (Renal and urinary disorders) | 0 | 0 | 1
Convulsion (Nervous system disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 1
Alcoholism (Psychiatric disorders) | 1 | 0 | 0
Schizophrenia, paranoid type (Psychiatric disorders) | 1 | 0 | 0
Schizophrenia (Psychiatric disorders) | 0 | 4 | 3
Paranoia (Psychiatric disorders) | 0 | 0 | 1
Psychotic disorder (Psychiatric disorders) | 0 | 0 | 1
Aggression (Psychiatric disorders) | 0 | 1 | 0
Agitation (Psychiatric disorders) | 0 | 1 | 0
Disturbance in social behavior (Psychiatric disorders) | 0 | 2 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 3 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Open- Label ALKS 3831 (N=255) | Olanzapine + Placebo (N=117) | ALKS 3831 (N=112)
Weight increased (Investigations) | 0 | 14 | 16
Alanine aminotransferase increased (Investigations) | 0 | 0 | 6
Nasopharyngitis (Infections and infestations) | 0 | 5 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Should an Investigator desire to disclose study results, Sponsor will review the results disclosure prior to public release and can embargo the disclosure for a period of at least 60 days. Revisions to the disclosure will be negotiated in good faith. For a multicenter study the Investigators agree to publish/publicly present the results together with the other sites for the 12 month period after study results are available unless Sponsor grants written permission in advance

DOCUMENTS (2):
  • Study Protocol (2016-03-01): https://cdn.clinicaltrials.gov/large-docs/18/NCT02161718/Prot_000.pdf
  • Statistical Analysis Plan (2017-01-20): https://cdn.clinicaltrials.gov/large-docs/18/NCT02161718/SAP_001.pdf